CLINICAL TRIAL: NCT04046393
Title: Chia Yi Chang Gung Memorial Hospital
Brief Title: Investigating the Effect of Herbal Medicine Nasal Irrigation on Treatment of Chronic Rhinitis and Sinusitis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201801970A3
Record Dates: First submitted 2019-08-05; First posted 2019-08-06 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Nasal Disease
Keywords: rhinitis, sinusitis, nasal irrigation, TCM
MeSH Terms: conditions — Nose Diseases; Rhinitis; Sinusitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Chinese Medicine(TCM) group (Experimental): nasal irrigation with Traditional herbal medicine(licorice) extract-saline isotonic solution
  Interventions: Device: Taiwan Scientific" noninvasive blood pressure meter TS-0411; Device: Meridian Energy Analysis Device(MEAD); Procedure: bacteria culture; Procedure: nasopharyngoscopic examination; Combination Product: TCM nasal irrigation
- Saline control group (Placebo Comparator): nasal irrigation with saline isotonic solution
  Interventions: Device: Taiwan Scientific" noninvasive blood pressure meter TS-0411; Device: Meridian Energy Analysis Device(MEAD); Procedure: bacteria culture; Procedure: nasopharyngoscopic examination

INTERVENTIONS:
Device: Taiwan Scientific" noninvasive blood pressure meter TS-0411 — measure autonomic nerve
Device: Meridian Energy Analysis Device(MEAD) — measure meridian energy
Procedure: bacteria culture — use culture swab to culture nasal discharge
Procedure: nasopharyngoscopic examination — use nasopharyngoscopy to determine the modified Lund-Kennedy endoscopic scoring system
Combination Product: TCM nasal irrigation — Chinese herbal medicine (licorice) extract solution with buffered salt packet and water in rinse bottle
  Arms: Traditional Chinese Medicine(TCM) group

SUMMARY:
This study investigate the nasal irrigation with Traditional herbal medicine extract-saline isotonic solution in the treatment of chronic rhinitis and sinusitis. Half of participants will receive Traditional herbal medicine extract-saline isotonic solution nasal irrigation, while the other half will receive saline alone nasal irrigation.

DETAILED DESCRIPTION:
In the program, the investigators plan to investigate a clinical triad to research the outcomes of nasal irrigation with Traditional herbal medicine extract-saline isotonic solution for treatment of chronic rhinitis and sinusitis. The aims of this study are listed below:

Aim 1: evaluating the outcomes and quality of life of nasal irrigation with Traditional herbal medicine extract-saline isotonic solution to treat enrolled patients with chronic rhinitis or sinusitis. The investigators use modern devices to evaluate the autonomic nerve, meridian energy and pulse. The questionnaires of quality of life and symptoms will be recorded. Nasal irrigation with saline alone will be conducted during the clinical triad to compare the effectiveness and quality of life with Traditional herbal medicine extract.

Aim 2: analyzing the changes of bacteria culture in nasal discharge collected during the clinical triad before and after nasal irrigation for investigating the microenvironment of Traditional herbal medicine extract-saline isotonic solution.

According to the research, the investigators will realize the improvement of using Traditional herbal medicine extract-saline isotonic solution for nasal irrigation to treat sino-nasal diseases, by investigating the changes of quality of life and microenvironment of nasal cavity. The nasopharyngoscopic examination, autonomic nerve, meridian energy and pulse were record to compare the effectiveness of Traditional herbal medicine extract-saline isotonic solution with nasal irrigation with saline alone.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnostic criteria for chronic rhinitis and sinusitis male and female volunteers.
2. Stop using oral and topical steroid and anti-histamine treatments >2 weeks prior to enrollment.
3. >20 years of age.

Exclusion Criteria:

1. Allergy to herbal medicine.
2. Presence of a sinus tumor.
3. Significant immune dysfunction.
4. Pregnancy and breast-feeding women.
5. Undergone nasal surgery <1 week prior to enrollment.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2019-12-31 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2022-02-14 (Estimated)

PRIMARY OUTCOMES:
WHOQOL-brief score (Taiwan version) | one month
  consisting of 28 items, each scored from 1 to 5; total score recorded as the sum of all items change from baseline: the questionnaires of quality of life

SECONDARY OUTCOMES:
22-item Sino-Nasal Outcome Test score (SNOT-22) | one month
  consisting of 22 items, each scored from 0 to 5; total score recorded as the sum of all items, 0 to 110 change from baseline: the questionnaires of chronic sinusitis severity
Total symptom score(TSS） | one month
  consisting of 4 items, each scored from 0 to 3; total score recorded as the sum of all items, 0 to 12 change from baseline: the questionnaires of chronic rhinitis severity
Autonomic nerve (HRV) | one month
  Low frequency (ms2), High frequency (ms2), LF/HF(indicate autonomic function) change from baseline
Meridian energy | one month
  Yang energy and Yin energy change from baseline
Posttreatment culture negativity | one month
  negative" means if no bacterial pathogen is identified on posttreatment culture but at least one has been present on pretreatment culture
Nasopharyngoscopic examination change | one month
  consisting of 3 items, each scored from 0 to 2; total score recorded as the sum of both side all items, 0 to 12 change from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Rung Yang, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Chiayi City, Taiwan